CLINICAL TRIAL: NCT04860011
Title: Sodium Glucose Cotransporter-2 Inhibitor DAPAgliflozin Versus Thiazide Diuretic in Patients With Heart Failure and Diuretic RESISTance: a Multi-centre, Open-label, Randomised Controlled Clinical Trial
Brief Title: DAPAgliflozin Versus Thiazide Diuretic in Patients With Heart Failure and Diuretic RESISTance
Acronym: DAPARESIST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN19CA407
Record Dates: First submitted 2021-04-06; First posted 2021-04-26 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — dapagliflozin; Metolazone

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, active-comparator, multi-centre, open label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SGLT2i (Experimental): Sodium-glucose Co-transporter-2 inhibitors
  Interventions: Drug: Dapagliflozin 10 MG Oral Tablet
- Thiazide (Experimental): Thiazide or thiazide like diuretic
  Interventions: Drug: Metolazone Tablets

INTERVENTIONS:
Drug: Dapagliflozin 10 MG Oral Tablet — Dapagliflozin 10mg once daily
  Other Names: dapagliflozin
  Arms: SGLT2i
Drug: Metolazone Tablets — Metolazone 5MG or 10MG once daily
  Other Names: metolazone
  Arms: Thiazide

SUMMARY:
To assess the effect of dapagliflozin compared with metolazone, added to furosemide, on diuresis and decongestion in hospitalised heart failure patients with diuretic resistance, and renal impairment. The primary analysis will be in patients with HFrEF but patients with HFpEF will also be recruited in an ancillary study and included in supplementary analyses.

DETAILED DESCRIPTION:
The investigators aim to assess whether SGLT2i (in addition to IV loop diuretic) results in greater diuresis and decongestion compared to the standard practice of treatment with the thiazide-like diuretic metolazone (in addition to IV loop diuretic) in patients hospitalised for heart failure, with both renal impairment and diuretic resistance. Dapagliflozin has received National Institute for Health and Care Excellence (NICE) approval as an add-on option to optimised standard care in patients with HFrEF. The investigators primary focus is patients with HFrEF as it is in ambulatory patients with this phenotype that SGLT2 inhibition has already been shown to reduce morbidity and mortality (DAPA-HF).However, the investigators will also enrol patients with HFpEF in an ancillary study as they present the same management challenges as patients with HFrEF and the study hypothesis and aims are as clinically relevant in HFpEF as in HFrEF. HFpEF patients in the ancillary study will undergo the same protocol as the main study. One recent trial demonstrating benefit of a SGLT1/2 inhibitor, the Effect of Sotagliflozin on Cardiovascular Events in Patients With Type 2 Diabetes Post Worsening Heart Failure (SOLOIST-WHF), included patients with both HFrEF and HFpEF hospitalised with worsening heart failure (NCT03521934). This trial demonstrated similar efficacy of sotagliflozin on cardiovascular death and worsening heart failure in patients with a LVEF <50% and ≥50%.There are other large trials currently underway specifically with SGLT2i in ambulatory patients with HFpEF underway. These trials are either fully recruited, or close to full enrolment. Both already have extensive follow-up of several thousand patients and are due to complete follow up in the next 1-2 years (EMPEROR-Preserved and DELIVER). Therefore, the findings will be contemporaneous and complementary to the results of those trials.

ELIGIBILITY:
Inclusion Criteria:

- Male or female ≥18 years of age

* Informed consent
* Primary reason for admission to hospital is worsening HF meeting the European Society of Cardiology (ESC) definition.14
* Diuretic Resistance as defined as: Lack of weight loss or absence of a negative fluid balance (as defined above) over the preceding 24 hours despite treatment with high dose IV loop diuretic (equivalent of ≥160mg IV furosemide in 24 hours)
* Plasma BNP ≥ 100 pg/mL or plasma NT-proBNP ≥ 400 pg/mL in current hospital admission
* eGFR <60 ml/min/1.73m2 required within 24 hours before randomisation
* Ongoing clinical evidence of congestion: pitting peripheral oedema and/or ascites and/or elevated jugular venous pressure, and/or radiographic or ultrasonic evidence of pulmonary congestion
* Expected hospital length of stay >3 days

Exclusion Criteria:

* Inability to give informed consent e.g. due to significant cognitive impairment

  * Intravascular volume depletion based on investigator's clinical assessment
  * eGFR <20 mL/min/1.73 m2
  * Alternative explanation for worsening renal function such as obstructive nephropathy, contrast induced nephropathy, or acute tubular necrosis
  * Enrollment in another randomised clinical trial involving medical or device-based interventions (co-enrolment in observational studies is permitted)
  * Women of child-bearing potential
  * History of allergy to SGLT2i or thiazide or thiazide-like diuretics or any of the excipients
  * Hypertrophic obstructive cardiomyopathy (HOCM) or significant valvular disease in whom surgical or percutaneous repair or replacement may be considered.
  * SGLT2i, thiazide or thiazide-like diuretics administration in the previous 48 hours prior to randomisation
  * Active genital tract infections
  * Anyone who, in the investigators' opinion, is not suitable to participate in the trial for other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-04-03 (Estimated)

PRIMARY OUTCOMES:
Diuretic effect | from randomisation to 48 hours
  Diuretic effect, as assessed by mean change in weight
Diuretic effect | from randomisation to 72 hours
  Diuretic effect, as assessed by mean change in weight
Diuretic effect | from randomisation to 96 hours
  Diuretic effect, as assessed by mean change in weight

SECONDARY OUTCOMES:
Change in congestion measured by ultrasound | from randomisation to 48 hours
  Change in congestion, assessed using lung ultrasound as a measure of the sum of B-lines across 8 zones
Change in congestion measured by ultrasound | from randomisation to 72 hours
  Change in congestion, assessed using lung ultrasound as a measure of the sum of B-lines across 8 zones
Change in congestion measured by ultrasound | from randomisation to 96 hours
  Change in congestion, assessed using lung ultrasound as a measure of the sum of B-lines across 8 zones
Loop diuretic efficiency | from randomisation to 48 hours
  Loop diuretic efficiency will be defined as weight loss in kilograms divided by furosemide equivalents in milligrams.
Loop diuretic efficiency | from randomisation to 72 hours
  Loop diuretic efficiency will be defined as weight loss in kilograms divided by furosemide equivalents in milligrams.
Loop diuretic efficiency | from randomisation to 96 hours
  Loop diuretic efficiency will be defined as weight loss in kilograms divided by furosemide equivalents in milligrams.
Change in ADVOR clinical congestion score | from randomisation to 48 hours
  Change in ADVOR clinical congestion score will be measured on a scale of 0 to 10 with 0 being the least congested
Change in ADVOR clinical congestion score | from randomisation to 72 hours
  Change in ADVOR clinical congestion score will be measured on a scale of 0 to 10 with 0 being the least congested
Change in ADVOR clinical congestion score | from randomisation to 96 hours
  Change in ADVOR clinical congestion score will be measured on a scale of 0 to 10 with 0 being the least congested

OTHER OUTCOMES:
Change in urinary spot sodium | from randomisation to 48 hours
  change in urinary spot urine measured in mmol/L
Change in urinary spot sodium | from randomisation to 72 hours
  change in urinary spot urine measured in mmol/L
Change in urinary spot sodium | from randomisation to 96 hours
  change in urinary spot urine measured in mmol/L
Change in NT-proBNP | from randomisation to 48 hours
  measured in pg/ml
Change in NT-proBNP | from randomisation to 72 hours
  measured in pg/ml
Change in NT-proBNP | from randomisation to 96 hours
  measured in pg/ml
Change in serum uric acid | from randomisation to 48 hours
  measured in umol/L
Change in serum uric acid | from randomisation to 72 hours
  measured in umol/L
Change in serum uric acid | from randomisation to 96 hours
  measured in umol/L
Serum uric acid ≥360 μmol/L | from randomisation to 48 hours
  measured in umol/L
Serum uric acid ≥360 μmol/L | from randomisation to 72 hours
  measured in umol/L
Serum uric acid ≥360 μmol/L | from randomisation to 96 hours
  measured in umol/L
Total net fluid loss | from randomisation to 48 hours
  difference between fluid intake and output measured in ml
Total net fluid loss | from randomisation to 72 hours
  difference between fluid intake and output measured in ml
Total net fluid loss | from randomisation to 96 hours
  difference between fluid intake and output measured in ml
Change in dyspnoea | from randomisation to 48 hours
  Change in dyspnoea (breathlessness) measured using a 7 point Likert scale (1= strong positive to 7 = strong negative) and a 11-point Dyspnoea Numerical Rating scale (0= not breathless at all to 10=breathlessness as bad as you can imagine)
Change in dyspnoea | from randomisation to 72 hours
  Change in dyspnoea (breathlessness) measured using a 7 point Likert scale (1= strong positive to 7 = strong negative) and a 11-point Dyspnoea Numerical Rating scale (0= not breathless at all to 10=breathlessness as bad as you can imagine)
Change in dyspnoea | from randomisation to 96 hours
  Change in dyspnoea (breathlessness) measured using a 7 point Likert scale (1= strong positive to 7 = strong negative) and a 11-point Dyspnoea Numerical Rating scale (0= not breathless at all to 10=breathlessness as bad as you can imagine)
Patient global assessment | from randomisation to 48 hours
  Change in patients perception of their own health measured using a 7 point Likert scale (1= strong positive to 7 = strong negative)
Patient global assessment | from randomisation to 72 hours
  Change in patients perception of their own health measured using a 7 point Likert scale (1= strong positive to 7 = strong negative)
Patient global assessment | from randomisation to 96 hours
  Change in patients perception of their own health measured using a 7 point Likert scale (1= strong positive to 7 = strong negative)
change in serum glucose | from randomisation to 72 hours
  measured in mmol/L
change in serum glucose | from randomisation to 48 hours
  measured in mmol/L
change in serum glucose | from randomisation to 96 hours
  measured in mmol/L
Time from randomisation to discharge | through study completion, an average of 5 days
  Time from randomisation to discharge measured in hours
In-hospital mortality | through study completion, an average of 5 days
  Number of patients who died in hospital
Rate of heart failure re-hospitalisation or death | through study completion (on average 5 days) and up to 90 days
  Number of patients who are re-admitted to hospital after initial discharge
Change in serum creatinine | from randomisation to 48 hours
  measured in umol/L
Change in serum creatinine | from randomisation to 72 hours
  measured in umol/L
Change in serum creatinine | from randomisation to 96 hours
  measured in umol/L
increase in serum creatinine concentration | from randomisation to 48 hours
  measured in umol/L
increase in serum creatinine concentration | from randomisation to 72 hours
  measured in umol/L
increase in serum creatinine concentration | from randomisation to 96 hours
  measured in umol/L
change in blood urea (nitrogen) | from randomisation to 48 hours
  measured in mmol/L
change in blood urea (nitrogen) | from randomisation to 72 hours
  measured in mmol/L
change in blood urea (nitrogen) | from randomisation to 96 hours
  measured in mmol/L
change in serum potassium | from randomisation to 48 hours
  measured in mmol/L
change in serum potassium | from randomisation to 72 hours
  measured in mmol/L
change in serum potassium | from randomisation to 96 hours
  measured in mmol/L
Serum potassium <3.5 mmol/L and ≥5.5 mmol/L | from randomisation to 48 hours
  measured in mmol/L
Serum potassium <3.5 mmol/L and ≥5.5 mmol/L | from randomisation to 72 hours
  measured in mmol/L
Serum potassium <3.5 mmol/L and ≥5.5 mmol/L | from randomisation to 96 hours
  measured in mmol/L
change in serum sodium | from randomisation to 48 hours
  measured in mmol/L
change in serum sodium | from randomisation to 72 hours
  measured in mmol/L
change in serum sodium | from randomisation to 96 hours
  measured in mmol/L
Serum sodium concentration <125 mmol/L | from randomisation to 48 hours
  measured in mmol/L
Serum sodium concentration <125 mmol/L | from randomisation to 72 hours
  measured in mmol/L
Serum sodium concentration <125 mmol/L | from randomisation to 96 hours
  measured in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: John McMurray, MBChB, Study Chair — University of Glasgow and NHS Greater Glasgow and Clyde
Locations (2):
- United Kingdom (2):
  - Glasgow Royal Infirmary, Glasgow, Strathclyde
  - Queen Elizabeth University Hospital, Glasgow, Strathclyde

IPD SHARING:
Plan to Share IPD: No
To be discussed and agreed at TSC

REFERENCES:
- [Derived] Yeoh SE, Osmanska J, Petrie MC, Brooksbank KJM, Clark AL, Docherty KF, Foley PWX, Guha K, Halliday CA, Jhund PS, Kalra PR, McKinley G, Lang NN, Lee MMY, McConnachie A, McDermott JJ, Platz E, Sartipy P, Seed A, Stanley B, Weir RAP, Welsh P, McMurray JJV, Campbell RT. Dapagliflozin vs. metolazone in heart failure resistant to loop diuretics. Eur Heart J. 2023 Aug 14;44(31):2966-2977. doi: 10.1093/eurheartj/ehad341. PMID 37210742